CLINICAL TRIAL: NCT04675606
Title: A Prospective Randomized Trial of Low Fiber Diet vs. Regular Diet in Postoperative Colorectal Patients With Ileostomies
Brief Title: Implementing a Low Fiber Diet vs. Regular Diet in Postoperative Colorectal Patients With Ileostomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Associate Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000894
Record Dates: First submitted 2020-12-02; First posted 2020-12-19 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Ileostomy; Complications; Bowel Obstruction; Postoperative Ileus
Keywords: Ileostomy; Bowel obstruction; Postoperative ileus; Low fiber diet; Regular diet
MeSH Terms: conditions — Intestinal Obstruction | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fiber diet (Active Comparator): Patients in this arm will receive low fiber diet starting postoperative day 1. This is currently the standard protocol at our institution.
  Interventions: Behavioral: Low fiber diet
- Regular diet (Experimental): Patients in this arm will receive regular diet starting postoperative day 1. This will be the experimental arm.
  Interventions: Behavioral: Regular diet

INTERVENTIONS:
Behavioral: Regular diet — Patients in the regular diet arm (which is the experimental arm) will not have any diet limitations and will be recommended to consume a healthy balanced diet for American adults as recommended by the United States Department of Agriculture (USDA) and US Food and Drug Administration (FDA).
  Arms: Regular diet
Behavioral: Low fiber diet — Patients in the low fiber diet arm (which is the control arm) will be recommended to consume foods that are low in fiber content per United Ostomy Associations of America Recommendations
  Other Names: Low residue diet
  Arms: Low fiber diet

SUMMARY:
The primary objective of this study is to prospectively evaluate rate of post-operative ileus or obstruction in patients with ileostomies receiving low fiber diet vs. regular diet starting post-operative day 1. The secondary objectives of this study are to compare the 30-day and 90-day readmission rates, length of stay, rate of high stoma output or need for antidiarrheals within 90 days, nausea score, level of pain, and overall quality of life amongst the patients studied.

DETAILED DESCRIPTION:
The proposed study is a prospective randomized study to compare two post-operative diets

1. Low fiber diet
2. Regular diet in patients undergoing elective or urgent colorectal surgery resulting in a loop or end ileostomy. The primary outcome measure is rate of post-operative ileus or obstruction in patients with ileostomies. The secondary objectives of this study are to compare the length of stay, 30-day and 90-day readmission rates, rate of high stoma output requiring antidiarrheal medication, nausea score, pain score, and overall quality of life amongst the patients studied.

All groups will be counseled and asked to consent for the study at the time of their preoperative clinic visit and copy of the protocol will be provided to them. Patients undergoing urgent surgery will be counseled and consented at the time decision for surgery is made. All groups will be started on either low fiber diet or regular diet on postoperative day 1. Of note, it is important to note that at our institution, a "low fiber diet" is equivalent to a "low residue diet" in our electronic medical records system. All groups will be assessed and examined daily, where nausea score and pain score will be recorded. Prior to discharge, both groups will receive consultation with a wound-ostomy care nurse who will perform ostomy teaching as well as diet/nutritional counseling. Patients in the low fiber diet arm will receive nutritional counseling advising that they follow a low fiber diet. Patients in the regular diet arm will receive nutritional counseling advising that they continue to follow a regular diet.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Undergoing elective or urgent major laparoscopic or open colorectal procedure resulting in new loop or end ileostomy creation
3. Urgent colorectal surgery is defined as operations performed during the same hospital admission, but greater than 24hrs after decision for surgery is made. Patients undergoing urgent colorectal surgery are not expected to require intensive care unit (ICU) admission postoperatively.
4. Willingness and ability to sign an informed consent document
5. No allergies to anesthetic or antiemetic
6. ASA physical status Class I - III
7. Aged 18-90 years

Exclusion Criteria:

1. Refusal to participate in the study
2. Undergoing emergent colorectal surgery. Emergent colorectal surgery is defined as patients who require immediate surgery < 24hrs after initial decision for surgery is made
3. Patients expected to require intensive care unit (ICU) admission postoperatively
4. Age <18 or > 90 years
5. Pregnancy
6. Patient with preoperative short-bowel syndrome or proximal stomas (jejunostomy)
7. Patients on preoperative total parenteral nutrition not expected to immediately commence postoperative enteral nutrition
8. Patients maintained NPO for any reason after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative ileus and obstruction | 90 days postoperatively
  evaluate rate of post-operative ileus or obstruction in patients with ileostomies receiving low fiber diet vs. regular diet starting post-operative day 1.

SECONDARY OUTCOMES:
Hospital readmission rates | 90 days postoperatively
  Hospital readmission rates
Hospital length of stay | Up to 90 days postoperatively
  Hospital length of stay
Volume of stoma output | 90 days postoperatively
  Average daily volume of stoma output
Need for antidiarrheal use | 90 days postoperatively
  Need for antidiarrheal use
Average maximum daily nausea score | 90 days postoperatively
  Average maximum daily nausea score on a scale of 0 to 2. A score of 0 means no presence of nausea, 1 denotes presence of nausea, and 2 denotes presence of vomiting. A higher score up to a maximum of 2 means a worse outcome compared to a lower score.
Average maximum daily pain score | 90 days postoperatively
  Average maximum daily pain score on a scale of 0 to 10. A score of 0 means a patient has no pain. A higher score up to the maximum of 10 means a worse outcome.
Quality of life | 90 days postoperatively
  Quality of life assessed using the Gastrointestinal Quality of Life Index (GIQLI) questionnaire. The GIQLI questionnaire has 36 items, each item is scored 0 to 4. The GIQLI has a range of 0 to 144. Higher score up to a maximum of 144 means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin SR, Wong YN, Uzzo RG, Beck JR, Egleston BL. Why Summary Comorbidity Measures Such As the Charlson Comorbidity Index and Elixhauser Score Work. Med Care. 2015 Sep;53(9):e65-72. doi: 10.1097/MLR.0b013e318297429c. PMID 23703645
- [Background] Chapman SJ, Pericleous A, Downey C, Jayne DG. Postoperative ileus following major colorectal surgery. Br J Surg. 2018 Jun;105(7):797-810. doi: 10.1002/bjs.10781. Epub 2018 Feb 22. PMID 29469195
- [Background] Correia MI, da Silva RG. The impact of early nutrition on metabolic response and postoperative ileus. Curr Opin Clin Nutr Metab Care. 2004 Sep;7(5):577-83. doi: 10.1097/00075197-200409000-00011. PMID 15295279
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Feo CV, Romanini B, Sortini D, Ragazzi R, Zamboni P, Pansini GC, Liboni A. Early oral feeding after colorectal resection: a randomized controlled study. ANZ J Surg. 2004 May;74(5):298-301. doi: 10.1111/j.1445-1433.2004.02985.x. PMID 15144242
- [Background] Levenstein S, Prantera C, Luzi C, D'Ubaldi A. Low residue or normal diet in Crohn's disease: a prospective controlled study in Italian patients. Gut. 1985 Oct;26(10):989-93. doi: 10.1136/gut.26.10.989. PMID 2996991
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Ray S, Mehta NN, Mangla V, Lalwani S, Mehrotra S, Chugh P, Yadav A, Nundy S. A Comparison Between the Comprehensive Complication Index and the Clavien-Dindo Grading as a Measure of Postoperative Outcome in Patients Undergoing Gastrointestinal Surgery-A Prospective Study. J Surg Res. 2019 Dec;244:417-424. doi: 10.1016/j.jss.2019.06.093. Epub 2019 Jul 18. PMID 31326707
- [Background] Reissman P, Teoh TA, Cohen SM, Weiss EG, Nogueras JJ, Wexner SD. Is early oral feeding safe after elective colorectal surgery? A prospective randomized trial. Ann Surg. 1995 Jul;222(1):73-7. doi: 10.1097/00000658-199507000-00012. PMID 7618972
- [Background] Wood T, Aarts MA, Okrainec A, Pearsall E, Victor JC, McKenzie M, Rotstein O, McLeod RS; iERAS group. Emergency Room Visits and Readmissions Following Implementation of an Enhanced Recovery After Surgery (iERAS) Program. J Gastrointest Surg. 2018 Feb;22(2):259-266. doi: 10.1007/s11605-017-3555-2. Epub 2017 Sep 15. PMID 28916971
- See also: Related Info — https://www.sealedenvelope.com/power/binary-noninferior/